CLINICAL TRIAL: NCT05845268
Title: Total Neoadjuvant Therapy Combined With Tislelizumab for Local Advanced Phase II Randomized Controlled Clinical Study of Middle and Low Rectal Cancer
Brief Title: Total Neoadjuvant Therapy Combined With Tislelizumab for Local Advanced of Middle and Low Rectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BFH-TNT-LARC
Record Dates: First submitted 2023-03-30; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2022-10

CONDITIONS: Locally Advanced Rectal Cancer
Keywords: neoadjuvant; Tislelizumab; PD-1; chemoradiation; LARC; randomized; controlled
MeSH Terms: interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Masking Description: Masking is not practically possible
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CRT+concurrent PD-1 inhibition (Experimental): Long-course chemoradiation plus PD-1 inhibition (Tislelizumab 200mg, 3 times, 3-week interval) starting on Day 8 of radiation therapy. TME surgery is scheduled in 10~13 weeks after completion of radiation.
  Interventions: Combination Product: Long-course chemoradiation, with Tislelizumab (PD-1 inhibitor)
- CRT without PD-1 inhibition (Active Comparator): Long-course chemoradiation plus PD-1 inhibition with no PD-1 inhibition. TME surgery is scheduled in 10~13 weeks after completion of radiation.
  Interventions: Combination Product: Long-course chemoradiation, without Tislelizumab (PD-1 inhibitor)

INTERVENTIONS:
Combination Product: Long-course chemoradiation, with Tislelizumab (PD-1 inhibitor) — Tislelizumab was added to long-course chemoradiotherapy (CRT) in LARC patients, CRT + concurrent tislelizumab was used in the Experimental arm, and CRT was used in the Active Comparator arm.
  Arms: CRT+concurrent PD-1 inhibition
Combination Product: Long-course chemoradiation, without Tislelizumab (PD-1 inhibitor) — Tislelizumab was added to long-course chemoradiotherapy (CRT) in LARC patients, CRT + concurrent tislelizumab was used in the Experimental arm, and CRT was used in the Active Comparator arm.
  Arms: CRT without PD-1 inhibition

SUMMARY:
This study is a prospective, randomized, open, controlled, multi-center phase II clinical trial, which included patients with locally advanced low rectal cancer as the research object, and evaluated the application of long-term concurrent chemoradiotherapy combined with tislelizumab versus long-term synchronous Efficacy and safety of chemotherapy and radiotherapy as neoadjuvant therapy for patients with locally advanced rectal cancer. The main endpoints of the study were clinical complete response (cCR) (including imaging and endoscopic complete response) and pathological complete response (pathological complete response, pCR). Secondary study endpoints are primary pathological response rate (MPR), objective response rate (ORR), disease-free survival (DFS), overall survival (OS), organ preservation rate (OPR), rectal cancer neoadjuvant therapy score (NAR ), quality of life score (QoL), safety and tolerability. They will be randomly divided into an experimental group (tislelizumab combined with long-term concurrent chemoradiotherapy) and a control group (long-term concurrent chemoradiotherapy) at a ratio of 2:1. Random stratification factors: 1. TNM stage (II/III); 2. Distance from the tumor to the anal verge (≥5cm, <5cm).

DETAILED DESCRIPTION:
This study plans to recruit 102 patients, aged 18-75 years old, male or female; rectal adenocarcinoma confirmed by histopathology; clinical stage II-III assessed by MRI (according to AJCC 8th edition); Margin ≤ 10 cm; surgical resection is possible.All patients should have no history of immune diseases, nor history of immunotherapy or radiotherapy. Eligible participants will be randomly assigned to Experiment Arm (50.4Gy radiation, capecitabine, and anti-PD1 starting at Day 8 of radiation) and Control Arm (50.4Gy radiation, capecitabine) in a 2：1ratio.

ELIGIBILITY:
Inclusion Criteria:

* Patients have been fully aware of the content of this study and signed the informed consent voluntarily;
* Patients with rectal cancers must satisfied all the following conditions:Stage II/III LARC (cT3-4aN0M0 and cT1-4aN1-2M0);Tumor distal location ≤ 10 cm from anal verge (MRI diagnosed);
* Patients regardless of gender with aged ≥18 years and ECOG score of 0 or 1;
* Physical and viscera function of patients can withstand major abdominal surgery;
* Patients are willing and able to follow the study protocol during the study;
* Patients give consent to the use of blood and pathological specimens for study;
* Within 28 days prior to enrolment, we must confirm a negative serological pregnancy test for child-bearing age women and they agree to use effective contraception for the duration of drug use and for 60 days after the last dose.

Exclusion Criteria:

* Patients have a present or previous active malignancy except the diagnosis of rectal cancer this time;
* Patients underwent major surgery within 4 weeks prior to study treatment;
* Patients have any condition affects the absorption of capecitabine through gastrointestinal tract;
* Patients have severe uncontrolled recurrent infections, or other severe uncontrolled concomitant diseases;
* Patients who are allergic to any of the ingredients under study;
* Patients with severe concomitant diseases with estimated survival ≤ 5 years;
* Patients with present or previous moderate or severe liver and kidney damage presently or previously;
* Patients have received other study medications or any immunotherapy currently or in the past;
* Patients preparing for or previously received organ or bone marrow transplant;
* Patients who received immunosuppressive or systemic hormone therapy for immunosuppressive purposes within 1 month prior to the initiation of study therapy;
* Patients with congenital or acquired immune deficiency (such as HIV infection);
* If patients with a history of uncontrolled epilepsy, central nervous system disease or mental disorder, the investigator will determine whether the clinical severity prevents the signing of informed consent or affects the patient's oral medication compliance;
* Patients with other factors that may affect the study results or cause the study to be terminated midway, such as alcoholism, drug abuse, other serious diseases (including mental illness) requiring combined treatment and severe laboratory examination abnormalities.
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
pCR rate | within 10 days after surgery
  pathological complete response rate
cCR rate | 12-13 weeks after radiotherapy ends
  clinical complete response rate

SECONDARY OUTCOMES:
NAR score | within 10 days after surgery
  Neoadjuvant rectal（NAR）score：It is based on the scoring criteria of preoperative treatment downstaging. The range is 0-201.46, with higher scores indicating worse prognosis.
OPR | immediately after surgery
  organ preservation rate
ORR | within 10 days after surgery
  objective response rate
immune-related adverse event rate | up to 30th day after surgery
  adverse event rate that is deemed to be associated with PD-1 inhibition

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Zhongtao, Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Export of individual patient data is a sensitive issue according to current Chinese laws